CLINICAL TRIAL: NCT02853240
Title: Transversal Monocentric Study of the Anatomophysiological Effect of Botulinum Toxin on the Spastic Muscle of Children With Cerebral Palsy
Brief Title: Effect of Botulinum Toxin on Muscles of Children With Cerebral Palsy
Acronym: TOXIMUS_CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL15_0540; 2016-001610-24 (EudraCT Number)
Record Dates: First submitted 2016-07-19; First posted 2016-08-02 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; children; muscle spasticity; botulinum toxin injection
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children with spastic CP receiving toxin injections (Experimental): Children with spastic cerebral palsy receiving toxin injections
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — A biopsy (specifically done for the study) of a muscle that has already been injected with botulinum toxin before inclusion of the patient in the study will be performed, taken during a planned surgery (for tendon transfer or muscle lengthening). A biopsy of a muscle that has never been injected with botulinum toxin may be performed during surgery. No biopsy will be made on a member that would not require surgery. Thus sampling will be conducted on a muscle requiring a surgery: 2 to 3 millimeters will be taken on 10 mm muscle before transfer or lengthening.

SUMMARY:
Cerebral palsy (CP) is a group of non-progressive motor dysfunction but often changing, secondary to injury or brain abnormalities that occur in early stages of development. In children with CP, the brain injury lead to a delayed motor development in the first weeks, associated with muscular spasticity. Drug treatments include oral treatments (baclofen and tizanidine) and injectable treatments like Botox (intramuscular injection) and neurolysis with alcohol or phenol (local injection into the nerve).

Regarding botulinum toxin, there is no study questioning its effectiveness. However, no publication on the pathophysiology of human muscle of the CP child after toxin injection was found. The action of the toxin on the neuromuscular junction (NMJ) and muscle structure is unknown in children with CP.

The primary objective of this study is to describe structural abnormalities of the CP child's muscle following multiple toxin injections in terms of NMJ fragmentation and axonal sprouting.

Secondary objectives:

To evaluate the relationship between:

* The severity of the motor impairment and muscle structural abnormalities.
* The clinical measure of spasticity and muscle structural abnormalities.
* To compare the structure spastic muscles with toxin injections and spastic muscle without toxin injections

For muscles with multiple toxin injections, assessing the relationship between :

* The number of toxin injections and muscle structural abnormalities.
* The date of the first injection and muscle structural abnormalities.
* The total dose of injected toxin in the muscle and its structural abnormalities.
* The nature of the product injected in the muscle and its structural abnormalities.

This innovative study will improve the knowledge on the effects of long-term botulinum toxin injections on the muscle (and therefore its safety in usual care), on the spastic muscle NMJ of CP children, on the pathophysiology of the CP child's muscle.

All the visits all acts will be performed according to usual patient follow-up. Only a biopsy will be performed in addition, taken from an injected muscle during a planned operation. A biopsy may also be performed on a muscle without toxin injection if the act is made possible by the planned surgery. No biopsy will be made on a muscle that would not require surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age Children > 7 years and <18 years
* With spastic cerebral palsy (all grades of the combined GMFCS
* Having an orthopedic surgical indication already planned on the lower limbs
* Receiving toxin injections
* With social security coverage
* Whose parents / holders of parental authority have signed the consent form

Exclusion Criteria:

* Patients with an evolutive CP
* Children with a baclofen pump
* Children who underwent neurotomy or functional dorsal rhizotomy, or alcohol or phenol injections

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Presence of neuromuscular junctions fragmentation (both qualitative and quantitative). | 6 months maximum (time of surgery)
  The biopsy is performed at the same time of a scheduled general anesthesia surgery (multisite surgery). The biopsy is 2 to 3 mm x 10 mm. It is a simple and quick gesture, usually practiced by surgeon
Presence of axonal sprouting (qualitative). | 6 months maximum (time of surgery)

SECONDARY OUTCOMES:
Proportion of muscles with neuromuscular junctions fragmentation (both qualitative and quantitative) and/or axonal sprouting (qualitative) according to patient's GMFCS grade (1 to 5). | 6 months maximum (time of surgery)
  The Gross Motor Function Classification System (GMFCS) is a 5 level clinical classification system that describes the gross motor function of people with cerebral palsy on the basis of self-initiated movement abilities.
Proportion of muscles with neuromuscular junctions fragmentation (both qualitative and quantitative) and/or axonal sprouting (qualitative) according to Ashworth score. | 6 months maximum (time of surgery)
  The Ashworth scale is bedside tool for assessing muscle spasticity in patients with neurological conditions. Ashworth grades as follows: 0, 1, 1+, 2, 3, 4.
Proportion of muscles with neuromuscular junctions fragmentation (both qualitative and quantitative) and/or axonal sprouting (qualitative) according to Tardieu score. | 6 months maximum (time of surgery)
  The Tardieu Scale is bedside tool for assessing muscle spasticity in patients with neurological conditions. Tardieu scale grades from 0 to 5.
Proportion of muscles with neuromuscular junctions fragmentation (both qualitative and quantitative) and/or axonal sprouting (qualitative) according to the number of toxin injections in the muscle. | 6 months maximum (time of surgery)
Proportion of muscles with neuromuscular junctions fragmentation (both qualitative and quantitative) and/or axonal sprouting (qualitative) according to the delay (in months) since the first toxin injection in the muscle | 6 months maximum (time of surgery)
Proportion of muscles with neuromuscular junctions fragmentation (both qualitative and quantitative) and/or axonal sprouting (qualitative) according to the total volume (IU) of injected toxin since the first injection in the muscle. | 6 months maximum (time of surgery)
Proportion of muscles with neuromuscular junctions fragmentation (both qualitative and quantitative) and/or axonal sprouting (qualitative) according to the brand of the injected toxin (Botox® or Dysport®). | 6 months maximum (time of surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No